CLINICAL TRIAL: NCT06813768
Title: Trattamento Delle Fistole Rettovaginali Di Crohn Mediante Combinazine Di Plug in Matrice Di Collagene (SURGIMEND®) Ed Infiltrazione Locale Di Tessuto Adiposo Autologo Microfratturato (LIPOGEMS®)
Brief Title: Treatment of Rectovaginal Crohn's Fistula by Combination of TAAM Injection and Biological Plug Placement
Acronym: LIPOPLUG
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Study currently suspended due to device-related issues
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LIPOPLUG - CROHN
Record Dates: First submitted 2025-01-28; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2024-12

CONDITIONS: Rectovaginal Fistula; Crohn Disease
Keywords: MICROFTACTURED ADIPOSE TISSUE; BIOLOGIC MESH; ENDOANAL FLAP; LIPOSUCTION
MeSH Terms: conditions — Rectovaginal Fistula; Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Randomization procedures and statistical analyses will be performed by an investigator not involved in the clinical evaluation or surgical treatment of patients. All clinical evaluations will be performed by independent co-investigators not involved in the surgical procedures and blinded to patient assignment. The dedicated radiologist who will evaluate the MRI scans will be blind to patient allocation. Surgeons will not be able to share information about the treatment used in the surgical procedure and will not be able to participate in any clinical evaluation of the MPC during the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Microfractured adipose tissue injection and plug placement (Experimental): Liposuction (up to 100 cc of adipose tissue) Processing of adipose tissue with lipogems system Drainage of sepsis, courettage of fistula tract Placement of biological prosthesis in the fistula tract, suturing the mesh with interrupted PDS sutures at the internal sphincter Injection of 15 cc of microfractured adipose tissue into the submucosa around the internal orifice and along the fistula tract
  Interventions: Device: Microfractured adipose tissue injection and plug placement
- endoanal mucosa flap (Active Comparator): A 6-0 absorbable suture will be placed on the skin at the level of the thigh to simulate liposuction Drainage of sepsis, courettage of fistula tract A U-shaped or vertical endoanal mucous flap will be made, after infiltration with 1:100,000 adrenaline of the mucosa surrounding the internal orifice, mobilization of the mucous flap, closure of the internal orifice at the muscular level with 2-0 absorbable stitches of PDS and suture of the mucosal flap with 3-0 absorbable vycril sutures.
  Interventions: Device: Microfractured adipose tissue injection and plug placement

INTERVENTIONS:
Device: Microfractured adipose tissue injection and plug placement — surgery + infiltration of micro-fractured autologous adipose tissue at the level of the internal orifice and placement of a biological prosthesis
  Other Names: Lipogems LGD 60 CND V0599 - RDM 1256088; Surgimend AWR 3X3 cm, 606-001-012 DM 409689/R

SUMMARY:
Interventional, prospective, randomized, controlled, double blind, parallel groups, nonprofit, single center trial

DETAILED DESCRIPTION:
The goal of this clinical trial is to compare, the efficacy of

* circumferential infiltration of microfractured autologous adipose tissue combined with the placement of a biological prosthesis in the fistula tract versus
* endoanal mucosal flap in terms of clinical and radiological healing (combined remission)

in patients with Crohn's rectovaginal fistulas refractory to standard treatment,

Secondary objectives are improvement of the clinical outcome (clinical remission, clinical response, failure), time elapsed between surgery and clinical outcome, onset of any recurrences, safety and improvement in quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed Crohn's disease
* presence of recto-vaginal fistula refractory to standard treatment (surgical drainage of sepsis and treatment with biological drg for at least 12 months)
* The patient has received, understood and signed the informed consent to actively participate in the study.
* The patient is able to understand the conditions of the study and to participate for the whole duration.

Exclusion Criteria:

* presence of oostomy
* Patients with active HIV, hepatitis C (HCV), hepatitis B (HBV), tuberculosis or other uncontrolled septic conditions.
* Patients who present technical difficulties, in the opinion of the investigator, in safely recovering the amount of adipose tissue necessary for the procedure.
* Patients with abdominal localization of Crohn's disease who may require general surgery during the study.
* Patients with active oncological or lymphoproliferative diseases
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients with recto-vaginal fistulas
Enrollment: 3 (Actual)
Dates: Start 2023-01-07 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
combined remission | 24 weeks
  clinical (absence of gas and/or fecal and/or purulent vaginal drainage after gentle digital compression) and radiological (absence of abscesses > 3 mm) closure of the fistula

SECONDARY OUTCOMES:
clinical remission | 12, 16, 20, 24 weeks
  absence of gas and/or fecal and/or purulent vaginal drainage after gentle digital compression) with radiological presence of abscesses > 3 mm
clinical response | 12, 16, 20, 24 weeks
  at least 50% reduction in drainage of the treated vaginal orifice that was draining at baseline despite gentle digital compression.
failure | 12, 16, 20, 24 weeks
  "no change/worsening" of vaginal drainage and patients who, in the judgment of the investigator, require treatment with antibiotics to control recurrent perianal sepsis
IBDQ score (quality of life) | 4, 8, 12, 16, 20, 24 weeks
  changes of Inflammatory Bowel Disease Questionnaire (IBDQ) scores
Incidence of adverse events | 4, 8, 12, 16, 20, 24 weeks
  comparison of incidence of adverse events and serious adverse events in the two arms

CONTACTS AND LOCATIONS:
Overall Officials: Silvio Laureti, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: Undecided